CLINICAL TRIAL: NCT04273438
Title: Determining the Clinical Utility of Using Virtual Reality Headsets to Assess Visual Function in Those With Glaucoma.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Queen's University, Belfast (Other)
Collaborators: University of Sussex (Other)
Responsible Party: Principal Investigator, Ruth Hogg, Principal Investigator, Queen's University, Belfast
Other Study IDs: 16/NI/0251
Record Dates: First submitted 2019-08-12; First posted 2020-02-18 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Glaucoma
Keywords: Perimetry; Virtual Reality; Visual field testing
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Visual field testing using Oculus Rift and Humphrey Visual Field Perimeter — Glaucoma patients at Queen's University, Belfast, will be invited to undergo both Visual field testing using the Oculus Rift and the gold-standard Humphrey 24-2 (Carl Zeiss Meditec, Dublin, CA) at two visits, and evaluating consistency for detecting visual field impairments.
Device: Visual Field Testing using HUmphrey 24-3 Perimeter — Glaucoma patients at Queen's University, Belfast, will be invited to undergo both Visual field testing using the Oculus Rift and the gold-standard Humphrey 24-2 (Carl Zeiss Meditec, Dublin, CA) at two visits, and evaluating consistency for detecting visual field impairments.

SUMMARY:
To validate a new virtual reality (VR) based visual field test against the gold standard clinical perimetry test (Humphrey Visual field test 24-2).

DETAILED DESCRIPTION:
Perimetry (or visual field testing) is a vision test used to evaluate a patient's peripheral vision. It involves a patient fixating on a central target and pressing a button when they see a spot of light in their peripheral vision. It is an important way of deciding whether Glaucoma is progressing or not. Next generation virtual reality (VR) technologies offer an exciting new way of conducting perimetry in either a clinical or home environment, allowing more affordable and more frequent monitoring of disease progression in glaucoma, and an easier and more comfortable experience for patients. The investigators propose to create a perimetry test using a commercially available head mounted display for VR, and to assess its accuracy in glaucoma patients in relation to standard automated perimetry.

ELIGIBILITY:
Inclusion Criteria:

- Patients with a clinical diagnosis of glaucoma with repeatable defects on standard automated perimetry.

Exclusion Criteria:

* Presence of other ocular disease which impacts vision such as age-related macular degeneration or diabetic retinopathy.
* Any physical limitation that would make the participant unable to place their head in the head-rest to perform Humphrey Perimetry (Eg some patients with arthritic or neck problems are unable to use the headrests of ophthalmic devices).
* Any cognitive impairment that would limit their ability to perform perimetry or a history of vertigo/dizziness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Professor Azuara-Blanco will identify participants who meet the criteria from his NHS clinics at the Shankill Health and Well-being Centre. He is part of both the direct care team and also a co-investigator on this application. Opportunistic sampling will be used to ensure that different severity levels of visual field deficit will be represented within the sample. Identification of potential participants will involve reviewing their patient records.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
mean deviation (MD) | All statisitcal analysis will take place once all data collection has ended, average 1 year..
  Mean deviation in decibels (dB), this is a standard summary measure generated by all perimetric tests and is considered to represent generalised loss of visual function.
Pattern Standard Deviation | All statisitcal analysis will take place once all data collection has ended, average 1 year..
  Pattern standard deviation in decibels (dB), this is a standard summary measure generated by all perimetric tests and is considered to represent localised loss of visual function.

SECONDARY OUTCOMES:
Repeatbility of both devices | All statisitcal analysis will take place once all data collection has ended, average 1 year..
  Bland and Altman plots and intra-class correlation coefficients will be generated for both tests for visit 1 vs visit 2 data.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth E Hogg, PhD, Principal Investigator — Queen's University, Belfast
Locations (1):
- NI Clinical Research Facility, Belfast, Northern Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-09): https://cdn.clinicaltrials.gov/large-docs/38/NCT04273438/Prot_SAP_000.pdf